CLINICAL TRIAL: NCT05043688
Title: Camrelizumab Plus Neoadjuvant Chemotherapy or Chemoradiotherapy Versus Neoadjuvant Chemoradiotherapy Alone for Resectable Locally Advanced Esophageal Squamous Cell Carcinoma (NICE 2): a Multi-center, Randomized Phase II Trial
Brief Title: Camrelizumab Plus Neoadjuvant Chemotherapy or Chemoradiotherapy Versus Chemoradiotherapy in Resectable ESCC.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhigang Li (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Zhigang Li, chief physician, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LS2160
Record Dates: First submitted 2021-09-05; First posted 2021-09-14 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Resectable Esophageal Squamous Cell Carcinoma
MeSH Terms: interventions — camrelizumab; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neoadjuvant Chemotherapy With Camrelizumab (Experimental): Chemotherapy: Paclitaxel（Albumin Bound）100mg/m2, Day 1,8,15，Carboplatin AUC=5mg/ml/min, Day 1； Camrelizumab: Day 1, every 3 weeks, 2 cycles; Postoperative adjuvant treatment: Camrelizumab maintenance
  Interventions: Drug: Camrelizumab
- Neoadjuvant Radiochemotherapy With Camrelizumab (Experimental): Chemotherapy: Paclitaxel 50mg/m2, Day 1,8,15,22,29，Carboplatin AUC=2mg/ml/min，Day 1,8,15,22,29 Camrelizumab: 200mg，Day 1,22 Radiotherapy: 41.4 Gy , D1-5/W Postoperative adjuvant treatment：Camrelizumab maintenance
  Interventions: Drug: Camrelizumab; Radiation: radiotherapy
- Neoadjuvant Radiochemotherapy (Active Comparator): Chemotherapy: Paclitaxel 50mg/m2, Day 1,8,15,22,29，Carboplatin AUC=2mg/ml/min，Day 1,8,15,22,29 Radiotherapy：41.4 Gy , D1-5/W. Postoperative adjuvant treatment: non-pCR: Camrelizumab maintenance; PCR: surveillance
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Drug: Camrelizumab — The study perform preoperative neoadjuvant therapy, surgery and postoperative adjuvant therapy on subjects. Preoperative neoadjuvant therapy includes 3 groups: iCamrelizumab combined with neoadjuvant chemotherapy; Camrelizumab combined with neoadjuvant radiochemotherapy, and neoadjuvant radiochemotherapy.
  Arms: Neoadjuvant Chemotherapy With Camrelizumab; Neoadjuvant Radiochemotherapy With Camrelizumab
Radiation: radiotherapy — The study perform preoperative neoadjuvant therapy, surgery and postoperative adjuvant therapy on subjects. Preoperative neoadjuvant therapy includes 3 groups: iCamrelizumab combined with neoadjuvant chemotherapy; Camrelizumab combined with neoadjuvant radiochemotherapy, and neoadjuvant radiochemotherapy.
  Arms: Neoadjuvant Radiochemotherapy; Neoadjuvant Radiochemotherapy With Camrelizumab

SUMMARY:
The purpose of this study is to explore the effectiveness and safety of neoadjuvant immune combined chemotherapy or radiochemotherapy compared with traditional neoadjuvant radiochemotherapy in patients with locally advanced Esophageal Squamous Cell Carcinoma.

DETAILED DESCRIPTION:
This study aimed to evaluate the efficacy and safety of adding immunotherapy to neoadjuvant chemotherapy (CT) or chemoradiotherapy (CRT) compared to neoadjuvant CRT alone for resectable locally advanced esophageal squamous cell carcinoma (ESCC)

ELIGIBILITY:
Inclusion Criteria:

1. The result of pathological biopsy showed esophageal squamous cell carcinoma;
2. Have not received systemic or local treatment for esophageal cancer in the past;
3. Age 18-75 years (including 18 and 75 years old), both male and female;
4. ECOG score 0-1;
5. Thoracic esophageal cancer assessed by CT/MRI/PET-CT etc. as resectable and the clinical stage is T1b-3N1-3M0 or T3N0M0, according to the 8th edition of AJCC staging;
6. Those who are expected to achieve R0 resection;
7. Voluntarily sign an informed consent form before treatment;
8. Plan to receive surgical treatment after neoadjuvant treatment is completed;
9. No surgical contraindications;
10. Normal function of major organs
11. Female subjects with fertility must undergo a serum pregnancy test within 72 hours before starting the study drug administration, and the result is negative, and take effective contraception during the trial and at least 3 months after the last administration Measures (such as intrauterine devices, contraceptives, or condoms); for male subjects whose partners are females of childbearing age, effective contraceptive measures should be taken during the trial and within 3 months after the last administration;
12. The subjects have good compliance and can follow up the efficacy and adverse events/reactions according to the requirements of the plan;

Exclusion Criteria:

1. There are unresectable factors, including unresectable tumors, unresectable contraindications for surgery, or rejection of surgery;
2. Patients with supraclavicular lymph node metastasis;
3. Poor nutritional status, BMI <18.5 Kg/m2; if the symptomatic nutritional support is corrected before randomization, the main investigator can continue to consider it after evaluation;
4. Those who are known to have a history of allergies to the drug components of this program;
5. Have received or are receiving any of the following treatments in the past:

   1. Any radiotherapy, chemotherapy or other anti-tumor drugs for tumors;
   2. Immunosuppressive drugs or systemic hormone drugs are being used within 2 weeks before the first use of the study drug to achieve immunosuppressive purposes (dose>10mg/day prednisone or equivalent dose); if there is no active autoimmune disease In the case of inhalation or topical use of steroids and prednisone doses> 10 mg/day or equivalent doses of adrenal cortex hormone replacement are allowed;
   3. Received a live attenuated vaccine within 4 weeks before using the study drug for the first time;
   4. Have undergone major surgery or severe trauma within 4 weeks before using the study drug for the first time;
6. A history of immunodeficiency, including a positive HIV test, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation or allogeneic bone marrow transplantation;
7. There are clinical symptoms or diseases of the heart that are not well controlled;
8. Severe infections (CTCAE v5.0> level 2) occurred within 4 weeks before the first use of the study drug, such as severe pneumonia, bacteremia, infectious comorbidities that require hospitalization, etc.; baseline chest imaging examinations suggest activity Pulmonary inflammation, symptoms and signs of infection in the 14 days before the first use of the study drug, or those who require oral or intravenous antibiotic treatment, except for the prophylactic use of antibiotics;
9. Participated in other drug clinical studies within 4 weeks before randomization;
10. People who are currently accompanied by interstitial pneumonia or interstitial lung disease, or have a history of interstitial pneumonia or interstitial lung disease that requires hormone therapy, or have other pulmonary fibrosis that may interfere with the judgment and management of immune-related lung toxicity , Organizing pneumonia (such as bronchiolitis obliterans), pneumoconiosis, drug-related pneumonia, idiopathic pneumonia, or subjects whose CT shows active pneumonia or severe lung dysfunction during the screening period; active tuberculosis;
11. Patients with any active autoimmune diseases or history of autoimmune diseases with the possibility of recurrence; patients with skin diseases that do not require systemic treatment, such as leukoplakia, psoriasis, hair loss, and insulin treatment Patients with controllable type I diabetes or a history of asthma, but who have been completely relieved during childhood without any intervention can be included in the group; patients with asthma who need bronchodilator intervention cannot be included in the group;
12. There is active hepatitis B (HBV-DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (hepatitis C antibody is positive, and HCV-RNA is higher than the lower limit of the analytical method);
13. Other malignant tumors have been diagnosed within 5 years before the first use of the study drug, unless malignant tumors with low risk of metastasis or death (5-year survival rate> 90%), such as fully treated skin basal cell carcinoma or squamous cell Skin cancer or cervical carcinoma in situ, etc., may be considered for inclusion;
14. Women who are pregnant or breastfeeding;
15. According to the judgment of the investigator, there are other factors that may lead to the forced termination of the study, such as suffering from other serious diseases (including mental illness) requiring combined treatment, alcoholism, drug abuse, family or social factors, which may affect the subjects Factors of safety or compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
EFS assessed by the investigator according to RECIST 1.1 | median EFS approximately over 45 months
  defined as event free survival,defined as the time from randomization to the occurrence of tumor progression/recurrence /death, whichever comes first

SECONDARY OUTCOMES:
OS | median OS approximately over 80 months
  defined as the time from registration to death due to any cause, or censored at date last known alive
R0 resection rate | within 28 working days after surgery
  defined as complete surgery resection rate
DFS | median DFS approximately over 40 months
  defined as the time from the date of surgery who completed R0 resection to local or distant recurrence, or death due to any cause, whichever occurs first;
HRQoL | approximately 48 months
  defined as quality and nutrition assessment
pCR | within 28 working days after surgery
  pCR is defined as pathological complete response(ypT0/TisN0)
MPR | within 28 working days after surgery
  MPR is defined as the percentage of subjects with <10% residual tumor in the primary tumor site
Adverse events (AEs) | through study completion, assessed up to 50 months
  Incidence and grade (including serious adverse events [SAEs] and immune-related adverse events [irAEs]), determined according to the NCI-CTCAE 5.0 criteria

OTHER OUTCOMES:
biomarker testing | approximately 48 months
  explore the correlation between the expression of PD-L1 and outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yang, Principal Investigator — Shanghai Chest Hospital
Locations (5):
- China (5):
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Anyang Tumour Hospital, Anyang
  - Sun yat-sen University Cancer Center, Guangzhou
  - Anhui Provincial Hospital, Hefei
  - Zhongshan Hospital of Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang Y, Zhu L, Cheng Y, Liu Z, Cai X, Shao J, Zhang M, Liu J, Sun Y, Li Y, Yi J, Yu B, Jiang H, Chen H, Yang H, Tan L, Li Z. Three-arm phase II trial comparing camrelizumab plus chemotherapy versus camrelizumab plus chemoradiation versus chemoradiation as preoperative treatment for locally advanced esophageal squamous cell carcinoma (NICE-2 Study). BMC Cancer. 2022 May 6;22(1):506. doi: 10.1186/s12885-022-09573-6. PMID 35524205
- See also: ClinicalTrials.gov Results Data Element Definitions for Interventional and Observational Studies (相关术语定义) — http://prsinfo.clinicaltrials.gov/results_definitions.html
- See also: Checklists, templates, and examples to help gather information needed to report results to ClinicalTrials.gov (试验结果填写指南) — http://prsinfo.clinicaltrials.gov/results_table_layout/ResultSimpleForms.html